CLINICAL TRIAL: NCT07090434
Title: Effect of an mHealth-based Digital Intervention to Support Multimodal Treatment in Patients With Fibromyalgia.
Brief Title: Effect of Bei App for Fibromyalgia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Madrid (Other)
Collaborators: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Raúl Ferrer-Peña, Dr, Universidad Autonoma de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: BEI.APP
Record Dates: First submitted 2025-07-02; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Fibromyalgia (FM)
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Psychoeducation program + mobile app (Experimental): In addition to the psychoeducation program (12 weekly group sessions, each lasting one hour), participants will receive access to the BEI mobile app, designed to reinforce education and exercise strategies outside clinical sessions. Participants will be instructed to use the app daily, guided by a to-do list including:
  * 1 educational module (interactive format) + 3 questions self-exam
  * 1 physical activity (video-guided, adapted by fatigue and pain level)
  * 1 gamified cognitive task (for memory, attention, speed processing and/or executive function)
  * Daily mood and symptom check-in
  Bei integrates adaptive feedback based on usage patterns, providing a more personalized experience to support long-term adherence.
  Interventions: Device: Mobile App + psychoeducation program
- Psychoeducation program alone (Active Comparator): Participants will attend 12 weekly group sessions, each lasting one hour, focused on psychoeducation. Sessions are delivered in person by trained professionals (physiotherapists and psychologists) from the association.
  Interventions: Behavioral: Psychoeducation program

INTERVENTIONS:
Device: Mobile App + psychoeducation program — Participants will attend 12 weekly group sessions, each lasting one hour, focused on psychoeducation. In addition to that, participants will receive access to the BEI mobile app, designed to reinforce education and exercise strategies outside clinical sessions. Participants will be instructed to use the app daily, guided by a to-do list including:
  * 1 educational module (interactive format) + 3 questions self-exam
  * 1 physical activity (video-guided, adapted by fatigue and pain level)
  * 1 gamified cognitive task (for memory, attention, speed processing and/or executive function)
  * Daily mood and symptom check-in
  Other Names: mhealth
  Arms: Psychoeducation program + mobile app
Behavioral: Psychoeducation program — Participants will attend 12 weekly group sessions, each lasting one hour, focused on psychoeducation.
  Arms: Psychoeducation program alone

SUMMARY:
Background: Fibromyalgia (FM) is a complex, chronic condition characterized by widespread musculoskeletal pain, cognitive dysfunction, fatigue, and emotional comorbidities such as anxiety and depression. These symptoms severely impact daily functioning and quality of life. Although non-pharmacological strategies-such as therapeutic exercise and patient education-are recommended as first-line treatments, their implementation outside the clinical setting remains a challenge due to low adherence and lack of continuity. Objective: To evaluate the effectiveness of a digital health intervention-BEI app-as a complement to usual care in improving clinical and functional outcomes among patients with fibromyalgia. Methods: This is a randomized controlled trial (RCT) with two parallel arms (1:1 allocation). A total of 70 adult participants with fibromyalgia (diagnosed per ACR 2016 criteria) will be recruited through a patient association in Madrid, Spain. The control group will receive 12 weeks of standard, in-person treatment consisting of group-based education and physical activity. The experimental group will receive the same in-person program plus daily access to the BEI mobile application, which includes educational modules, physical and cognitive training, symptom tracking, and personalized feedback. Outcomes will be assessed at baseline, week 6 (mid-intervention), week 12 (post-intervention), and week 24 (follow-up). Primary outcomes include pain intensity (VAS) and functional impact (FIQR). Secondary outcomes include catastrophizing, self-efficacy, cognitive function, physical activity, anxiety, depression, quality of life, app engagement, and satisfaction. Expected results: The results of this trial will provide evidence regarding the potential of mHealth tools to enhance adherence, self-efficacy, and functional outcomes in individuals with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be adults between 18 and 65 years of age with a clinical diagnosis of fibromyalgia according to the 2016 criteria established by the American College of Rheumatology (ACR).
* All participants must be actively enrolled in the group sessions offered by the patient association and possess the ability to use a smartphone or tablet compatible with the BEI app.
* Informed consent must be provided voluntarily.
* Additionally, participants are required to have a minimum level of digital health literacy, operationalized as a score equal to or greater than 2.5 in at least four dimensions of the eHealth Literacy Questionnaire (eHLQ).

Exclusion Criteria:

* Participants will be excluded if they present with severe or unstable psychiatric disorders, such as schizophrenia or uncontrolled major depression.
* Other exclusion criteria include medical comorbidities that contraindicate physical activity, current pregnancy, or concurrent participation in another digital health program or the use of similar therapeutic applications.
* Individuals with cognitive impairments or technological limitations that prevent the use of the app or participation in digital assessments will also be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-01-07 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | Baseline (week 0) - half treatment (week 6) - end of the treatment (week 12) - follow up (week 24)
  Pain intensity will be measured using a 100 mm Numeric Rating Scale (NRS), where 0 represents "no pain" and 100 represents the "worst pain imaginable." Participants will mark a point on the line that best reflected the pain they were experiencing at the time of measurement. Higher scores indicated higher levels of pain, and the administration required less than one minute
Functional Impact | Baseline (week 0) - half treatment (week 6) - end of the treatment (week 12) - follow up (week 24)
  It will be measured using the Revised Fibromyalgia Impact Questionnaire (FIQR), a tool designed to assess the impact of fibromyalgia on patients' daily lives. The FIQR consists of 21 items that evaluate various dimensions, including physical functioning, symptom severity, general health, and pain perception. Items are scored on a scale from 0 to 10, with higher scores indicating a greater impact of the disease. It has demonstrated high internal consistency, with a Cronbach's alpha ranging from 0.91 to 0.95

SECONDARY OUTCOMES:
Pain Catastrophizing | Baseline (week 0) - half treatment (week 6) - end of the treatment (week 12) - follow up (week 24)
  It will be assessed using the Pain Catastrophizing Scale (PCS), which measures the tendency to think catastrophically about pain. The scale consists of 13 items covering three dimensions: rumination, magnification, and helplessness in the face of pain. A Likert scale from 0 to 4 is used, with higher scores indicating greater levels of catastrophizing. The PCS has demonstrated test-retest reliability of 0.84 and adequate internal consistency, with a Cronbach's alpha of 0.79
Self-Efficacy | Baseline (week 0) - half treatment (week 6) - end of the treatment (week 12) - follow up (week 24)
  it will be assessed using the Pain Self-Efficacy Questionnaire (PSEQ), a self-report questionnaire consisting of 10 items, designed to measure an individual's self-efficacy in managing pain. It assesses the patient's confidence in their ability to perform daily activities despite pain, reflecting their sense of control and autonomy in the face of painful situations. The PSEQ has demonstrated excellent internal consistency, with a Cronbach's alpha of 0.92, and high test-retest reliability with an ICC of 0.90
Cognitive Function | Baseline (week 0) - half treatment (week 6) - end of the treatment (week 12) - follow up (week 24)
  It will be measured using the Montreal Cognitive Assessment (MoCA), a screening tool designed to quickly assess cognitive function in adults. The MoCA consists of 30 items that evaluate various cognitive domains, including attention, memory, language, visuospatial abilities, and executive functions. The test takes approximately 10-15 minutes to complete and is particularly useful in both clinical and research settings for a rapid and effective evaluation of cognitive functioning. The MoCA has demonstrated good validity and reliability across various populations, with a Cronbach's alpha of 0.77 and an intra-rater correlation of 0.92
Physical Activity | Baseline (week 0) - half treatment (week 6) - end of the treatment (week 12) - follow up (week 24)
  it will be assessed using the International Physical Activity Questionnaire (IPAQ - short version), which is designed to quickly and efficiently measure physical activity levels in adults. It includes questions that evaluate the frequency and intensity of physical activities performed over the past week, including walking, moderate activity, and vigorous activity
Kinesiophobia | Baseline (week 0) - half treatment (week 6) - end of the treatment (week 12) - follow up (week 24)
  it will be assessed using a self-report The Tampa Scale for Kinesiophobia (TSK-11), a self-report questionnaire comprising 11 items. The internal consistency of the TSK is high, with Cronbach's alpha coefficients ranging from 0.74 to 0.93, indicating strong reliability. Test-retest reliability is also good, with correlation coefficients ranging from 0.75 to 0.88
Anxiety | Baseline (week 0) - half treatment (week 6) - end of the treatment (week 12) - follow up (week 24)
  it will be assessed using using the Anxiety subscale of the validated Spanish version of the Hospital Anxiety and Depression Scale (HADS), which is divided into two subscales of 7 items each: 1) Depression (HADS-Dep); and 2) Anxiety (HADS-Anx). The subscales of HADS showed internal consistency indices recommended for screening tools. The items in HADS demonstrated a positive correlation with the total score of the anxiety and depression subscales. HADS was found to perform well in assessing the symptom severity and caseness of anxiety disorders and depression in both somatic, psychiatric, and primary care patients and in the general population
Depression | Baseline (week 0) - half treatment (week 6) - end of the treatment (week 12) - follow up (week 24)
  it will be assessed using the Depression subscale of the validated Spanish version of the Hospital Anxiety and Depression Scale (HADS), which is divided into two subscales of 7 items each: 1) Depression (HADS-Dep); and 2) Anxiety (HADS-Anx). The subscales of HADS showed internal consistency indices recommended for screening tools. The items in HADS demonstrated a positive correlation with the total score of the anxiety and depression subscales. HADS was found to perform well in assessing the symptom severity and caseness of anxiety disorders and depression in both somatic, psychiatric, and primary care patients and in the general population
Quality of Life EQ-5D | Baseline (week 0) - half treatment (week 6) - end of the treatment (week 12) - follow up (week 24)
  it will be measured with the EuroQoL-5D (EQ-5D) questionnaire, a self-report instrument for assessing health-related quality of life. It comprises three elements: a descriptive scale of 5 factors, a second element composed of a vertical NRS, and a social value index generated by the instrument. The EQ-5D has shown good psychometric properties
Digital Literacy | Baseline (week 0)
  Using 4 dimensions of the eHLQ as a screening tool.
App Engagement: Frequency of App Use | final of the treatment (week 12) and follow up (24 week)
  Engagement with the app will be assessed by measuring the frequency of app use, defined as the number of distinct access sessions per week.
  Unit of Measure: Number of sessions per week
App Engagement: Session Length | final of the treatment (week 12) and follow up (24 week)
  Average duration of each session using the app will be recorded automatically. Unit of Measure: Minutes per session (mean)
App Engagement: Completion of Logs | final of the treatment (week 12) and follow up (24 week)
  Engagement will be measured by the proportion of daily symptom or activity logs completed by participants relative to the number expected during the intervention period.
  Unit of Measure: Percentage of logs completed (%)
App Engagement: Completion of Modules | final of the treatment (week 12) and follow up (24 week)
  Engagement with the educational component of the app will be measured by the proportion of completed modules relative to the total number available.
  Unit of Measure: Percentage of modules completed (%)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy concerns and data protection regulations. Although the data will be anonymized, the sensitivity of health-related information from participants with chronic pain conditions requires strict adherence to ethical standards and GDPR compliance. Therefore, no IPD will be made publicly available.